CLINICAL TRIAL: NCT02728245
Title: Randomized Phase 2 Trial Comparing Preoperative Dienogest Therapy Followed by Surgery vs. Upfront Surgery to Save Ovarian Reserve in Young Women With Ovarian Endometrioma
Brief Title: Trial Comparing Preoperative Dienogest Therapy Followed by Surgery vs. Upfront Surgery to Save Ovarian Reserve in Young Women With Ovarian Endometrioma
Acronym: DOROSY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Placebo cannot be prepared
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Korea University Guro Hospital (Other); Ajou University School of Medicine (Other); Ewha Womans University Mokdong Hospital (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kidong Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUBH_GO_052
Record Dates: First submitted 2016-03-19; First posted 2016-04-05 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Reserve; Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo drug 1 tablet per day will be prescribed for 3months before surgery in ovarian endometrioma patients.
  Dienogest(DNG) 2mg 1 tablet per day will be prescribed for 2 months from 1month after surgery.
  Interventions: Drug: Dienogest; Drug: Placebo drug; Procedure: Surgery
- Case group (Experimental): Dienogest(DNG) 2mg 1 tablet per day will be prescribed for 3months before surgery in ovarian endometrioma patients.
  Dienogest(DNG) 2mg 1 tablet per day will be prescribed for 2 months from 1month after surgery.
  Interventions: Drug: Dienogest; Procedure: Surgery

INTERVENTIONS:
Drug: Dienogest — Dienogest 2mg po qd
Drug: Placebo drug — Placebo 1 table po qd
  Arms: Control group
Procedure: Surgery — conservative surgery without intent to oophorectomy

SUMMARY:
Randomized phase 2 trial comparing preoperative dienogest therapy followed by surgery vs. upfront surgery to save ovarian reserve in young women with ovarian endometrioma

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ovarian endometrioma ≥ 5cm or bilateral ovarian endometriomas with any size diagnosed by ultrasonography.
* In Patients with previous unilateral salpingo-oophorectomy (USO)
* Unilateral ovarian endometrioma with any size is eligible
* 20 ≤ Age ≤ 45 and premenopause
* Plan to undergo conservative surgery for endometriomas

Exclusion Criteria:

* Pregnant women or women who were suspected to be pregnant
* Women with current venous thromboembolism or history of such diseases
* Women with current arterial disease or cardiovascular diseases (e.g. myocardial infarction, cerebrovascular diseases, or ischemic heart diseases) or history of such diseases
* Women with current diabetes with vascular lesions or history of such diseases
* Women with current severe liver diseases or history of severe liver diseases with abnormal liver function
* Women with current liver tumor or history of liver tumor
* Women with current or history of sex-hormone dependent malignant tumor or women who were suspected to have a sex-hormone dependent malignant tumor
* Women with vaginal bleeding of unknown causes
* Women with a history of allergic reaction to elements of DNG
* Women with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Women whose non-compliance is expected
* Lactation (treatment with DNG is not recommended in lactating women due to possible excretion in breast milk)
* Any medication that could result in an excessive accumulation, impaired metabolism, or altered excretion of the study drug or might interfere with the conduct of the study or the interpretation of the results

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Compare the mean change of serum Anti-Mullerian Hormone (AMH) level | 3 month after surgery

SECONDARY OUTCOMES:
Compare the mean change of serum AMH level | 1 month after surgery
Compare the trend of mean change of serum AMH level | 1 and 3 month after surgery
Compare the mean change of serum AMH level | baseline and after preoperative dienogest/placebo therapy for 3 months
Compare the revised American fertility society (AFS) score | At surgery
compare the surgical time (minute) | intraoperative
  surgical time (minute)
Brief Pain Inventory (BPI) scores | baseline, 1 month after surgery and 3 month after surgery
number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | All adverse events from randomization to postoperative 3 months
Mean change of diameter of endometrioma measured by ultrasonography after preoperative dienogest/placebo therapy for 3months | baseline and after preoperative dienogest/placebo therapy for 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No